CLINICAL TRIAL: NCT07283146
Title: The Effect of EX-PLISSIT Model-Based Sexual Counseling on Perceptions of Sexuality, Sexual Quality of Life, and Sexual Satisfaction in Postmenopausal Women
Brief Title: The Effect of EX-PLISSIT Model-Based Sexual Counseling in Postmenopausal Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NESLİHAN YILMAZ SEZER (Other)
Responsible Party: Sponsor-Investigator, NESLİHAN YILMAZ SEZER, Faculty of Nursing, Ankara University
Organization: Ankara University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 18/242
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Postmenopause

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Counseling Group (Experimental)
  Interventions: Other: EX-PLISSIT Model-Based Sexual Counseling
- Control Group (No Intervention)

INTERVENTIONS:
Other: EX-PLISSIT Model-Based Sexual Counseling — Women in the experimental group will receive sexual counseling based on the EX-PLISSIT model. The steps to be followed in accordance with this model are as follows:
  Session 1 Permission Limited Information Specific Suggestions IT - Intensive Therapy
  Session 2 At the beginning of the interview, the data collection forms will be re-administered, and the homework assigned in the first session will be discussed. The information needed by the woman, in line with her questions, will be provided within the steps of the EX-PLISSIT model: permission, limited information, specific suggestions, and, if necessary, intensive therapy. At the end of the second session, the women will be given an appointment for the final assessment to be conducted two months later.
  Session 3 At the beginning of the interview, the data collection forms will be administered for the last time, the woman's questions (if any) will be answered, and the session will be concluded.
  Arms: Counseling Group

SUMMARY:
The study will be conducted in two groups as counseling and control. Participants will be approached at the Public Education Center. After postmenopausal women are evaluated according to eligibility criteria, those who are eligible will be informed about the research and written informed consent will be obtained from those who agree. Random assignment of women to the study groups will be carried out using randomization.

This study aimed to determine the effects of sexual counseling based on the EX-PLISSIT model on sexual quality of life, sexual satisfaction, and perceptions of sexuality in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal, defined as having had no menstrual periods or vaginal bleeding in the last 12 months,
* Under 65 years of age,
* Married,
* Having entered menopause naturally,
* Able to understand, speak, and read Turkish.

Exclusion Criteria:

* Women with diagnosed conditions that may significantly affect sexual quality of life (such as diabetes, hypertension, heart disease, pulmonary diseases, cancer types, psychiatric disorders, or a history of neurological stroke),
* Women using medications known to negatively affect sexual function (including psychotropic drugs, cardiac and antihypertensive medications, anticonvulsants, opioids, antinarcotics, H2-receptor antagonists, and antihistamines),
* Those who have previously received or are currently receiving hormone replacement therapy,
* Those with a diagnosis of sexual dysfunction in themselves or their partners,
* Those who have experienced major stressful life events (such as an accident, trauma, or the death or severe illness of a close relative) within the three months prior to the study,
* Women with a serious impairment that affects their ability to complete data collection forms,
* Not willing to participate in the study.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-07-17 (Estimated); Study Completion 2026-07-17 (Estimated)

PRIMARY OUTCOMES:
Change in Sexual Life Quality | at the beginning of the study, 1 month later and 3 months later
  The scale is easy to apply, 6-point Likert type, which individuals can answer on their own, and consists of 18 items. Each item is expected to be answered considering the sexual life in the last four weeks. Each item of the scale is scored between 1 and 6. The items of the scale are scored as "I totally agree"=1, "I strongly agree"=2, "I partially agree"=3, "I partially disagree"=4, "I strongly disagree"=5, "I strongly disagree"=6 and 1 Questions 5, 9, 13 and 18 are reverse coded. The range of points that can be obtained from the scale is between 18-108.
Change in sexual satisfaction | at the beginning of the study, 1 month later and 3 months later
  VAS is a 10-cm-long measurement tool. The left end of the scale reads "I am not satisfied at all" and the right end reads "very satisfied". A high score on the scale indicated a high level of satisfied and a score of 0 pointed to no satisfied.
Change in sexuality perception | at the beginning of the study, 1 month later and 3 months later
  Sexuality Perception Scale in Menopause The 12-item, 5-point Likert-type scale consists of two subdimensions: Perceptions Restricting Sexuality and Perceptions Related to the Continuation of Sexual Life. The minimum possible score on the scale is 12, and the maximum score is 60. Higher scores indicate more positive perceptions regarding sexuality during menopause.

IPD SHARING:
Plan to Share IPD: No